CLINICAL TRIAL: NCT07000500
Title: INSIDE: Intervenção da Suplementação Nutricional na Melhoria do Declínio Cognitivo no Idoso.
Brief Title: INSIDE: Intervention in Nutritional Supplementation to Improve Cognitive Decline in Elderly.
Acronym: INSIDE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Paço (Other)
Responsible Party: Sponsor-Investigator, Maria Paço, PhD, Cooperativa de Ensino Superior, Politécnico e Universitário
Organization: Cooperativa de Ensino Superior, Politécnico e Universitário (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INSIDE_2025
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Dysfunction, Cognitive Disorder; Dietary Supplements
Keywords: Cognitive Decline; Mild Cognitive Impairment; Aging; Nutritional Supplementation
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Supplement (Experimental): Participants in this arm will receive a daily dose of a nutritional supplement for 90 consecutive days. The supplement is administered orally and aims to improve cognitive performance in older adults with signs of cognitive decline. Participants will also complete cognitive assessments before and after the intervention.
  Interventions: Dietary Supplement: Nutritional Supplement
- Placebo (Placebo Comparator): Participants in this arm will receive a daily dose of an inert placebo that matches the supplement in appearance, taken orally for 90 consecutive days. The placebo is used as a control to compare the effects of the nutritional supplement on cognitive performance. Participants will undergo the same cognitive assessments as the experimental group.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nutritional Supplement — Participants in this arm will receive a daily dose of a nutritional supplement for 90 consecutive days. The supplement is administered orally and aims to improve cognitive performance in older adults with signs of cognitive decline. Participants will also complete cognitive assessments before and after the intervention.
  Arms: Nutritional Supplement
Other: Placebo — Participants in this arm will receive a daily dose of an inert placebo that matches the supplement in appearance, taken orally for 90 consecutive days. The placebo is used as a control to compare the effects of the nutritional supplement on cognitive performance. Participants will undergo the same cognitive assessments as the experimental group.
  Arms: Placebo

SUMMARY:
This study investigates the effect of nutritional supplementation on cognitive performance in older adults over a 90-day period using a double-blind randomized controlled design. The study includes 50 participants, aged 65 or older, randomly assigned to either a supplement group or a placebo group. Participants will be randomly assigned to either the experimental or control group. Assessments will be conducted pre- and post-intervention to determine the effect of the supplementation on cognitive performance. Key outcomes include cognitive status measured by MoCA, adherence to supplementation, and potential side effects. The findings will provide insights into the potential role of nutritional interventions in mitigating age-related cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Community-dwelling adults aged 65 years or older Evidence of mild cognitive decline (score < 26 on the Montreal Cognitive Assessment - MoCA) Ability to provide written informed consent Willingness and ability to comply with study procedures and attend scheduled evaluations

- Exclusion Criteria: Diagnosis of dementia or any neurodegenerative disease (e.g., Alzheimer's, Parkinson's) Epilepsy and neurologically related conditions Severe sensory deficits (e.g., profound visual or hearing impairment) that impair cognitive assessment Current use of cognitive-enhancing medications or supplements that cannot be discontinued History of allergy or intolerance to components of the nutritional supplement Unstable chronic medical conditions (e.g., uncontrolled diabetes, heart failure, renal insufficiency) Participation in another clinical trial in the previous 3 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Cognitive Performance | baseline and 90 days
  Change in cognitive performance measured by MoCA before and after intervention (90 days)

SECONDARY OUTCOMES:
Adherence to supplementation protocol | Daily, from Day 1 to Day 90
  Adherence will be monitored through a participant-completed intake diary, in which each participant records daily supplement or placebo consumption over the 90-day period. Adherence will be calculated as the percentage of days with confirmed intake out of the total study period. High adherence is defined as ≥80% of doses taken.
Occurrence of adverse effects | Continuous, from baseline to Day 90
  Participants will be asked to report any physical or psychological symptoms that arise during the 90-day supplementation period. Data will be collected through structured interviews at the end of the study and verified against notes recorded in the daily intake diary. Symptoms will be classified according to severity (mild, moderate, severe) and suspected relation to the intervention.
Self-reported use of other supplements | Baseline and 90 days
  At baseline and at the end of the study, participants will complete a questionnaire about their regular use of other dietary supplements or medications. This information will help identify potential confounding factors related to cognitive performance.
Self-perceived quality of life | baseline and 90 days
  Quality of life will be assessed using a brief, validated self-report questionnaire (e.g., EQ-5D or WHOQOL), administered before and after the intervention. The tool measures domains such as physical health, mental well-being, and social functioning. Scores will be compared to evaluate potential changes associated with the intervention.
Depressive symptoms | Baseline and Day 90
  Symptoms of depression will be assessed using a short validated screening tool (e.g., Geriatric Depression Scale - short form) at baseline and post-intervention. The tool provides a numerical score that will be used to evaluate changes in depressive symptomatology throughout the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Saúde do Vale do Ave, Vila Nova de Famalicão, Braga District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
Deciding whether to share Individual Participant Data (IPD) involves weighing several considerations... we have to further reflect to make an informed decision about sharing IPD, balancing the potential benefits to the scientific community with the responsibility to protect participant rights and data integrity.